CLINICAL TRIAL: NCT04743167
Title: IVF Versus Surgery for the Treatment of Infertility Associated to Ovarian and Deep Peritoneal Endometriosis
Brief Title: IVF Versus Surgery for Endometriosis Related Infertility
Acronym: SVIDOE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: IRCCS San Raffaele (Other); ASST Fatebenefratelli Sacco (Other); Ministero della Salute, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENDO-2020-23670289
Record Dates: First submitted 2021-02-02; First posted 2021-02-08 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Endometriosis
Keywords: IVF; surgery; endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgery (Active Comparator): Patients undergoing surgery for endometriosis, after surgery, will receive indications for seeking for a natural pregnancy up to 12 months from the time of randomization
  Interventions: Procedure: Surgery
- In Vitro Fertilization (Active Comparator): Patients included in the IVF arm will undergo three complete cycles of IVF (i.e. three oocytes retrievals regardless of the number of embryo transfers)
  Interventions: Procedure: IVF

INTERVENTIONS:
Procedure: Surgery — Laparoscopic treatment of endometriotic lesions
  Arms: Surgery
Procedure: IVF — Up to three completed cycles of IVF
  Arms: In Vitro Fertilization

SUMMARY:
The management of endometriosis-related infertility remains controversial. In particular, there is an equipoise for infertile women with endometriotic lesions detected at ultrasound. These women can be managed with either surgery or in vitro fertilization (IVF). The two approaches radically differ and they have never been compared with a randomized trial. As a consequence, affected women currently receive contrasting information and the mode of treatment substantially differ among centres, reflecting the local expertise of physicians rather than clinical needs.

The present study aims at clarify whether IVF could be superior to surgery in infertile women with endometriotic lesions detected at ultrasound. This topic will be addressed comparing the two approaches in terms of effectiveness and cost-effectiveness. In addition, the study will disentangling whether the endometriosis-related systemic inflammatory mechanisms may have an impact on the quality of folliculogenesis and on IVF outcomes. This specific objective will be pursued through the characterization and analysis of circulating extracellular vesicles (EV)-immunologic, proteomic and miRNA signatures and measurement of steroid hormones in follicular fluid.

DETAILED DESCRIPTION:
Women accepting to enter the study will be randomized to either surgery and then natural pregnancy seeking or a program of three complete IVF cycles (i.e. three oocytes retrievals regardless of the number of embryo transfers performed). The initial time point will be the time of randomization. Women of both study groups will initiate treatment (surgery or IVF) in a shortest delay, maximum 3 months. Only live birth pregnancies and initiating within a 12-months period starting from this time point will be included in the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age < 40 years
* Pregnancy seeking for more than 12 months
* Regular menstrual cycle, i.e. mean cycle interval between 21 and 35 days
* Ultrasonographic diagnosis of ovarian endometriomas or deep peritoneal endometriosis.
* Normal seminal analysis based on WHO criteria
* Absence of ureteral stenosis or intestinal subocclusive symptoms

Exclusion Criteria:

* Previous surgery for endometriosis
* Previous IVF cycles
* Contraindication to pregnancy
* Hydrosalpinx
* Endometriomas with a mean diameter > 4 cm
* Submucosal fibroids or large intramural or subserosal fibroids (≥ 5 cm).
* Doubtful sonographic findings that do not allow to reliably rule out malignancy.
* Obstacles to regular sexual intercourses (sexual disturbances or logistic problems)

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 206 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Live birth rate from pregnancies started within 12 months since randomization | up to 12 months since randomization
  to assess whether IVF is more effective than surgery in obtaining a live birth and, if so, what is the magnitude of this benefit

SECONDARY OUTCOMES:
Cost-effectiveness evaluation of the two different approaches in the treatment of endometriosis | 12 months
  to assess whether or not IVF is more cost-effective than surgery. To this aim, costs will be calculated based on the local charges for treatments (Diagnostic-related groups) and the costs of drugs supported by the public health system. The perspective will be the one of the public health provider.
Detachment of inflammatory mediators that might interfere with IVF through analysis of extracellular vescicles (EV). | 3 months
  to understand whether the endometriosis-related systemic inflammatory milieu demonstrated by the presence of circulating EVs characterized by an inflammatory signature may influence the folliculogenesis quality and IVF outcomes. EVs will be assessed by: Nanoparticle Tracking analysis (NTA) to determine their total values and their distribution; specific markers for the various lymphocyte populations by flow cytometry to assess the immunological origin; miRNA profile and proteomic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Benaglia, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (3):
- Italy (3):
  - ASST-FBF-Sacco, Presidio Ospedaliero Macedonio Melloni, Milan, MI
  - IRCCS San Raffaele, Milan, MI
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, MI

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ottolina J, Vignali M, Papaleo E, Vigano P, Somigliana E, Ferrari S, Liprandi V, Belloni G, Reschini M, Candiani M, Vercellini P, Benaglia L. Surgery versus IVF for the treatment of infertility associated to ovarian and deep endometriosis (SVIDOE: Surgery Versus IVF for Deep and Ovarian Endometriosis). Clinical protocol for a multicenter randomized controlled trial. PLoS One. 2022 Aug 3;17(8):e0271173. doi: 10.1371/journal.pone.0271173. eCollection 2022. PMID 35921357